CLINICAL TRIAL: NCT04047693
Title: Efficacy and Safety of Neoadjuvant Chemotherapy With Dose Dense MVAC Followed by Radical Surgery in Patients With MIBC and Locally Advanced Urothelial Carcinoma of Bladder: Phase II, Single-arm Study
Brief Title: Neoadjuvant Dose Dense MVAC in MIBC and Locally Advanced Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwonoh Park, MD phD, Professor, clinical research, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ddMVAC
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Muscle Invasive Bladder Cancer; Urothelial Carcinoma; Neoadjuvant Chemotherapy
Keywords: dose dense MVAC; neoadjuvant chemotherapy; Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Prospective, Single institution, Open-label, Phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ddMVAC (Experimental): 4 cycles of neoadjuvant chemotherapy using dose dense MVAC with G-CSF
  Interventions: Drug: dose dense MVAC with pegylated GCSF

INTERVENTIONS:
Drug: dose dense MVAC with pegylated GCSF — Methotrexate, 30 mg/m2 IV bolus, Day 1 Vinblastine, 3 mg/m2 IV bolus, Day2 Doxorubicin, 30 mg/m2 IV bolus, Day2 Cisplatin, 70 mg/m2 IV over 1hr, Day2 Pegylated G-CSF, 6mg SC, Day 3 every 2 weeks

SUMMARY:
The objective is to investigate the efficacy and safety of four cycles of ddMVAC with G-CSF support in patients with MIBC and locally advanced UC

DETAILED DESCRIPTION:
* Currently, most treatment guidelines including NCCN recommend a neoadjuvant chemotherapy (NAC) as a standard of care in muscle invasive bladder cancer (MIBC).
* Although standard NAC regimen is controversial due to rare of head to head study between each regimens, cisplatin based multidrug combination regimens such as MVAC, GP, and dose dense MVAC (ddMVAC) with G-CSF supports are regarded as a backbone treatment on the basis of the results from previous studies.
* Application of NAC is still relatively slow adoption in real practice. These slow adoption result from intuitive concerns such as significant toxicity of multidrug combination chemotherapy represented by MVAC and delayed application of radical surgical treatment in non-responder
* The ddMVAC with G-CSF support regimen showed an improved efficacy compared with GP regimen, and tolerable compared with standard MVAC using application of routine G-CSF support and high intensity of cisplatin.
* In case of clinically lymph node evolvement (cN+) is not for strict NAC, but patient with cN+ UC have been treated induction chemotherapy of similar NAC regimens and surgical treatment. So, this study included MIBC plus cN+ UC as locally advanced UC.
* In Korea, there is a low adoption of NAC, additionally rare of ddMVAC with G-CFS in locally advanced UC. It is supposed concerns related with toxicity of ddMVAC. Although the concern is likely not true considering the previous result of the Western, there has not been studied ddMVAC as NAC in Asian including Korean.
* The objective of this trial is to assess the efficacy and safety of four cycles of ddMVAC with G-CSF support in patients with locally advanced UC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed urothelial cancer of bladder.
2. Locally advanced status for planning surgical treatment (Bladder, confirm muscle invasiveness using TURBT, or cT3-4a and N1-3 using imaging studies)
3. Age 18 years or older
4. Eastern Cooperative Oncology Group performance status 0-1
5. Adequate organ and bone marrow function for cisplatin based chemotherapy

   A. Adequate bone marrow function: Absolute Neutrophil Count (ANC) ≥ 1,500/µL, platelets ≥ 100,000/µL, hemoglobin ≥ 9 g/dL)

   B. Adequate renal function: creatinine < 1.5 x upper normal limit (UNL) or creatinine clearance(Ccr) using Cockroft and Gault formula ≥ 50 ml/min

   C. Adequate hepatic function: bilirubin < 1.5 x UNL, AST/ALT levels <5.0 x UNL, alkaline phosphatase < 5 x UNL (except in case of bone metastasis without any liver disease)
6. Women should use contraceptive medication for 6 months after the end of the study or she would be post-menopause status. Men should consent with the contraception for 6 months after the end of the study or he would be infertile.
7. Patients should sign a written informed consent before study entry.

Exclusion Criteria:

1. Histologic types other than urothelial cell carcinoma should be excluded. However, urothelial cell types combined with squamous or glandular features are allowed.
2. Excess of 4 weeks after initial imaging studies. But, allow the patients to enrollment of study if they is reassessed and reconfirm the localized status using subsequent imaging studies. In this case, clinical stage is decided as following imaging studies.
3. Prior systemic chemotherapy (But prior intravesical chemotherapy was allowed)
4. Peripheral sensory neuropathy grade 2 or worse according to NCI CTCAE
5. History of treatment with drugs of another clinical trial within 30 days before enrollment.
6. Concomitant severe medical, surgical, or psychiatric disease or problems which can affect the results of the clinical trial or have possibilities of unexpected medical problems caused be the drug of clinical trial

   A. Unstable angina, myocardial infarction, uncontrolled arrhythmias, symptomatic angina pectoris, cardiac failure within the previous 6 months

   B. Active infection which would compromise the patients

   C. Liver cirrohosis or chronic active hepatitis

   D. Poor pulmonary function (DLCO ≤ 50% of normal or resting O2 saturation ≤ 90%)

   E. Clinically significant hemoptysis or gastrointestinal bleeding within previous 6 months

   F. Major psychiatric disorders or other inadequate psychiatric problems according to the physicians decision
7. History of another malignancy (but treated malignancy at least two years before enrollment were allowed, and cured non-melanoma skin cancer, any cured in-situ carcinoma, clinically insignificant localized prostate cancer, or papillary thyroid carcinoma are allowed even diagnosed less than 2 years before enrollment).
8. Pregnant or lactating women, women of childbearing potential not employing adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic response | From date of enrollment until curative intended surgical treatment, assess up to 2 years
  No residual tumor (ypT0N0) and partial response (ypTis-1N0) in surgical specimen

SECONDARY OUTCOMES:
Rate of pathologic complete response (pCR rate) | From date of enrollment until curative intended surgical treatment, assess up to 2 years
  No residual tumor (ypT0N0) in surgical specimen
Overall survival (OS) | From date of enrollment until death, assess up to 3 years
  Time from enrollment until death from any cause
Event free survival (EFS) | From date of enrollment until death, assess up to 3 years
  Time from enrollment until the earliest occurrence of disease progression in inoperablity, locoregional recurrence, distant metastasis, or death from any cause
Adverse events related with ddMVAC | From date of enrollment until 8 weeks after last chemotherapy of ddMVAC
  Adverse events related with ddMVAC using CTCAE 4.0
Surgical treatment related complication | From surgical treatment until 60 the days after surgical treatment
  Surgical treatment related complication

CONTACTS AND LOCATIONS:
Overall Officials: Kwonoh Park, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Witjes JA, Comperat E, Cowan NC, De Santis M, Gakis G, Lebret T, Ribal MJ, Van der Heijden AG, Sherif A; European Association of Urology. EAU guidelines on muscle-invasive and metastatic bladder cancer: summary of the 2013 guidelines. Eur Urol. 2014 Apr;65(4):778-92. doi: 10.1016/j.eururo.2013.11.046. Epub 2013 Dec 12. PMID 24373477
- [Result] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Result] International Collaboration of Trialists; Medical Research Council Advanced Bladder Cancer Working Party (now the National Cancer Research Institute Bladder Cancer Clinical Studies Group); European Organisation for Research and Treatment of Cancer Genito-Urinary Tract Cancer Group; Australian Bladder Cancer Study Group; National Cancer Institute of Canada Clinical Trials Group; Finnbladder; Norwegian Bladder Cancer Study Group; Club Urologico Espanol de Tratamiento Oncologico Group; Griffiths G, Hall R, Sylvester R, Raghavan D, Parmar MK. International phase III trial assessing neoadjuvant cisplatin, methotrexate, and vinblastine chemotherapy for muscle-invasive bladder cancer: long-term results of the BA06 30894 trial. J Clin Oncol. 2011 Jun 1;29(16):2171-7. doi: 10.1200/JCO.2010.32.3139. Epub 2011 Apr 18. PMID 21502557
- [Result] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524
- [Result] Madersbacher S, Hochreiter W, Burkhard F, Thalmann GN, Danuser H, Markwalder R, Studer UE. Radical cystectomy for bladder cancer today--a homogeneous series without neoadjuvant therapy. J Clin Oncol. 2003 Feb 15;21(4):690-6. doi: 10.1200/JCO.2003.05.101. PMID 12586807
- [Result] Millikan R, Dinney C, Swanson D, Sweeney P, Ro JY, Smith TL, Williams D, Logothetis C. Integrated therapy for locally advanced bladder cancer: final report of a randomized trial of cystectomy plus adjuvant M-VAC versus cystectomy with both preoperative and postoperative M-VAC. J Clin Oncol. 2001 Oct 15;19(20):4005-13. doi: 10.1200/JCO.2001.19.20.4005. PMID 11600601
- [Result] Ho PL, Willis DL, Patil J, Xiao L, Williams SB, Melquist JJ, Tart K, Parikh S, Shah JB, Delacroix SE, Navai N, Siefker-Radtke A, Dinney CP, Pisters LL, Kamat AM. Outcome of patients with clinically node-positive bladder cancer undergoing consolidative surgery after preoperative chemotherapy: The M.D. Anderson Cancer Center Experience. Urol Oncol. 2016 Feb;34(2):59.e1-8. doi: 10.1016/j.urolonc.2015.08.012. Epub 2015 Oct 1. PMID 26421586
- [Result] Zargar-Shoshtari K, Zargar H, Lotan Y, Shah JB, van Rhijn BW, Daneshmand S, Spiess PE, Black PC. A Multi-Institutional Analysis of Outcomes of Patients with Clinically Node Positive Urothelial Bladder Cancer Treated with Induction Chemotherapy and Radical Cystectomy. J Urol. 2016 Jan;195(1):53-9. doi: 10.1016/j.juro.2015.07.085. Epub 2015 Jul 21. PMID 26205531
- [Result] Sweeney P, Millikan R, Donat M, Wood CG, Radtke AS, Pettaway CA, Grossman HB, Dinney CP, Swanson DA, Pisters LL. Is there a therapeutic role for post-chemotherapy retroperitoneal lymph node dissection in metastatic transitional cell carcinoma of the bladder? J Urol. 2003 Jun;169(6):2113-7. doi: 10.1097/01.ju.0000067601.29966.4a. PMID 12771730
- [Result] Reardon ZD, Patel SG, Zaid HB, Stimson CJ, Resnick MJ, Keegan KA, Barocas DA, Chang SS, Cookson MS. Trends in the use of perioperative chemotherapy for localized and locally advanced muscle-invasive bladder cancer: a sign of changing tides. Eur Urol. 2015 Jan;67(1):165-170. doi: 10.1016/j.eururo.2014.01.009. Epub 2014 Jan 23. PMID 24472710
- [Result] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Result] Yin M, Joshi M, Meijer RP, Glantz M, Holder S, Harvey HA, Kaag M, Fransen van de Putte EE, Horenblas S, Drabick JJ. Neoadjuvant Chemotherapy for Muscle-Invasive Bladder Cancer: A Systematic Review and Two-Step Meta-Analysis. Oncologist. 2016 Jun;21(6):708-15. doi: 10.1634/theoncologist.2015-0440. Epub 2016 Apr 6. PMID 27053504
- [Result] Zargar H, Espiritu PN, Fairey AS, Mertens LS, Dinney CP, Mir MC, Krabbe LM, Cookson MS, Jacobsen NE, Gandhi NM, Griffin J, Montgomery JS, Vasdev N, Yu EY, Youssef D, Xylinas E, Campain NJ, Kassouf W, Dall'Era MA, Seah JA, Ercole CE, Horenblas S, Sridhar SS, McGrath JS, Aning J, Shariat SF, Wright JL, Thorpe AC, Morgan TM, Holzbeierlein JM, Bivalacqua TJ, North S, Barocas DA, Lotan Y, Garcia JA, Stephenson AJ, Shah JB, van Rhijn BW, Daneshmand S, Spiess PE, Black PC. Multicenter assessment of neoadjuvant chemotherapy for muscle-invasive bladder cancer. Eur Urol. 2015 Feb;67(2):241-9. doi: 10.1016/j.eururo.2014.09.007. Epub 2014 Sep 23. PMID 25257030
- [Result] Sternberg CN, de Mulder PH, Schornagel JH, Theodore C, Fossa SD, van Oosterom AT, Witjes F, Spina M, van Groeningen CJ, de Balincourt C, Collette L; European Organization for Research and Treatment of Cancer Genitourinary Tract Cancer Cooperative Group. Randomized phase III trial of high-dose-intensity methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) chemotherapy and recombinant human granulocyte colony-stimulating factor versus classic MVAC in advanced urothelial tract tumors: European Organization for Research and Treatment of Cancer Protocol no. 30924. J Clin Oncol. 2001 May 15;19(10):2638-46. doi: 10.1200/JCO.2001.19.10.2638. PMID 11352955
- [Result] Plimack ER, Hoffman-Censits JH, Viterbo R, Trabulsi EJ, Ross EA, Greenberg RE, Chen DY, Lallas CD, Wong YN, Lin J, Kutikov A, Dotan E, Brennan TA, Palma N, Dulaimi E, Mehrazin R, Boorjian SA, Kelly WK, Uzzo RG, Hudes GR. Accelerated methotrexate, vinblastine, doxorubicin, and cisplatin is safe, effective, and efficient neoadjuvant treatment for muscle-invasive bladder cancer: results of a multicenter phase II study with molecular correlates of response and toxicity. J Clin Oncol. 2014 Jun 20;32(18):1895-901. doi: 10.1200/JCO.2013.53.2465. Epub 2014 May 12. PMID 24821881
- [Result] Choueiri TK, Jacobus S, Bellmunt J, Qu A, Appleman LJ, Tretter C, Bubley GJ, Stack EC, Signoretti S, Walsh M, Steele G, Hirsch M, Sweeney CJ, Taplin ME, Kibel AS, Krajewski KM, Kantoff PW, Ross RW, Rosenberg JE. Neoadjuvant dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin with pegfilgrastim support in muscle-invasive urothelial cancer: pathologic, radiologic, and biomarker correlates. J Clin Oncol. 2014 Jun 20;32(18):1889-94. doi: 10.1200/JCO.2013.52.4785. Epub 2014 May 12. PMID 24821883
- [Result] Zargar H, Shah JB, van de Putte EEF, Potvin KR, Zargar-Shoshtari K, van Rhijn BW, Daneshmand S, Holzbeierlein JM, Spiess PE, Winquist E, Horenblas S, Dinney C, Black PC, Kassouf W. Dose dense MVAC prior to radical cystectomy: a real-world experience. World J Urol. 2017 Nov;35(11):1729-1736. doi: 10.1007/s00345-017-2065-x. Epub 2017 Jun 17. PMID 28625005
- [Result] Zargar H, Shah JB, van Rhijn BW, Daneshmand S, Bivalacqua TJ, Spiess PE, Black PC, Kassouf W; Collaborators. Neoadjuvant Dose Dense MVAC versus Gemcitabine and Cisplatin in Patients with cT3-4aN0M0 Bladder Cancer Treated with Radical Cystectomy. J Urol. 2018 Jun;199(6):1452-1458. doi: 10.1016/j.juro.2017.12.062. Epub 2018 Jan 9. PMID 29329894
- [Result] Kitamura H, Tsukamoto T, Shibata T, Masumori N, Fujimoto H, Hirao Y, Fujimoto K, Kitamura Y, Tomita Y, Tobisu K, Niwakawa M, Naito S, Eto M, Kakehi Y; Urologic Oncology Study Group of the Japan Clinical Oncology Group. Randomised phase III study of neoadjuvant chemotherapy with methotrexate, doxorubicin, vinblastine and cisplatin followed by radical cystectomy compared with radical cystectomy alone for muscle-invasive bladder cancer: Japan Clinical Oncology Group Study JCOG0209. Ann Oncol. 2014 Jun;25(6):1192-8. doi: 10.1093/annonc/mdu126. Epub 2014 Mar 24. PMID 24669010